CLINICAL TRIAL: NCT05777785
Title: A Pilot Study to Assess the Efficacy and Safety of a Novel Device (VIZO Glasses) in the Management of ADHD in Adults
Brief Title: A Novel Device for the Management of ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIZO Specs Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIZO_003
Record Dates: First submitted 2023-02-15; First posted 2023-03-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: ADHD
Keywords: ADHD; Peripheral Retinal Stimulation; non-pharmacological
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): VIZO Glasses- personalized
  Interventions: Device: VIZO Glasses

INTERVENTIONS:
Device: VIZO Glasses — Eyeglasses with personalized peripheral retinal stimuli

SUMMARY:
This is a 2-months study, where eligible ADHD adult participants will be provided with personalized VIZO glasses.

DETAILED DESCRIPTION:
This study was designed as a pilot single-center, open-label study of 2 months treatment. Following the enrollment, the participants will go through an adjustment process where they will be fitted with a personalized pair of VIZO Glasses. The participants will be instructed to wear the glasses throughout the day for two months. A follow-up visit at the end of the 2-month treatment will be conducted to assess the efficacy of VIZO Glasses on managing ADHD symptoms, using the Conners Continuous Performance Test-3, the Adult ADHD Self-Report Scale (ASRS), Behavior Rating Inventory of Executive Function Adults (BRIEF-A), and Clinical Global Impression-Improvement (CGI-I) .

ELIGIBILITY:
Inclusion Criteria:

* Documented history of primary ADHD diagnosis by certified clinicians
* Age 18-40 y
* Written informed consent
* Able and willing to complete all required ratings and assessments

Exclusion criteria:

* Any current psychiatric / neurological comorbidity (e.g., epilepsy, Autism, depression, TBI, etc), other than ADHD
* ADHD Medications (stimulants, non-stimulants, other)
* Neurofeedback, cognitive training

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Elyoseph, PhD, Principal Investigator — Max Stern Academic College of Emek Yezreel
Locations (1):
- Max Stern Academic College of Emek Yezreel, Haifa, Israel

REFERENCES:
- [Derived] Richter Y, Gordon C, Vainstein G, Bublil-Mor C, Geisinger D, Meital-Kfir N, Elyoseph Z. A novel intervention for treating adults with ADHD using peripheral visual stimulation. Front Psychiatry. 2023 Oct 20;14:1280440. doi: 10.3389/fpsyt.2023.1280440. eCollection 2023. PMID 37928920

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 108 partcipants met the inclusion criteria. Two participants failed to comply with the personalization process due to difficulty staying awake or using a cell phone during the test, resulting in 106 participants receiving the intervention.
Groups:
- Active: VIZO Glasses- personalized
  VIZO Glasses: Eyeglasses with personalized peripheral retinal stimuli. Participants were instructed to wear the glasses throughout the day for two months.
Period: Overall Study
Arm/Group | Active
Started | 106
Completed | 100
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes all 100 participants who completed the study, excluding three participants that were excluded due to major protocol deviations.
Arm/Group | Active
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.51 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Adult ADHD Self-Report Scale (ASRS) - Total Score [Mean (Standard Deviation); unit: units on a scale] — The Adult ADHD Self-Report Scale (ASRS) is a self-report instrument that comprises eighteen items that correspond with the DSM-V-TR criteria for ADHD. Subjects are asked to rate 18 symptom items using a 5-point Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Total scores range from 0 to 72, based on the sum of all 18 questions. Higher scores mean more symptoms and higher ADHD's impairments. Lower values represent better outcomes.
  units on a scale | 39.76 (12.10)
Adult ADHD Self-Report Scale (ASRS) - Inattentiveness Subscale [Mean (Standard Deviation); unit: units on a scale] — The inattentiveness sub-scale of the ASRS measures difficulties with focusing on details, organisation, remembering appointments, making careless mistakes, and concentration. It includes 9 symptom items using a 5-point Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Total scores range from 0 to 36, based on the sum of all questions. Higher scores mean more symptoms and higher inattentiveness' impairments.
  units on a scale | 21.2 (6.68)
Adult ADHD Self-Report Scale (ASRS) - Hyperactivity/Impulsivity subscale [Mean (Standard Deviation); unit: units on a scale] — The Hyperactivity/Impulsivity subscale of the ASRS assesses two components of hyperactivity/impulsivity. Firstly it measures motor difficulties such as sitting still, staying seated, and ability to relax. It also measures verbal difficulties such as controlling talking, interrupting others, and waiting turns. It includes 9 symptom items using a 5-point Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Total scores range from 0 to 36, based on the sum of all questions. Higher scores mean more symptoms and higher inattentiveness' impairments.
  units on a scale | 18.56 (6.64)

OUTCOME MEASURES:

1. Primary Outcome: Adult ADHD Self-Report Scale (ASRS) - Total Score at Baseline and 2 Months Follow up
Description: The Adult ADHD Self-Report Scale (ASRS) is a self-report instrument that comprises eighteen items that correspond with the DSM-V-TR criteria for ADHD. Subjects are asked to rate 18 symptom items using a 5-point Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Total scores range from 0 to 72, based on the sum of all 18 questions. Higher scores mean more symptoms and higher ADHD's impairments. Lower values represent better outcomes. The ASRS has two subscales that can be used to identify ADHD subtypes - Inattentiveness and Hyperactivity/Impulsivity. Each subscale contains 9 questions.
Time Frame: Baseline, 2 months
Population: Two participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 95
score on a scale
  Baseline | 39.76 (1.24)
  End of study | 38.27 (1.31)

2. Primary Outcome: Adult ADHD Self-Report Scale (ASRS) - Inattentiveness Subscale Score at Baseline and 2 Months Follow up
Description: The inattentiveness sub-scale of the ASRS measures difficulties with focusing on details, organisation, remembering appointments, making careless mistakes, and concentration. It includes 9 symptom items using a 5-point Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Total scores range from 0 to 36, based on the sum of all questions. Higher scores mean more symptoms and higher inattentiveness' impairments.
Time Frame: Baseline, 2 months
Population: Two participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active
Number analyzed (Participants) | 95
score on a scale
  Baseline | 21.20 (0.69)
  End of study | 20.22 (0.72)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — Power analysis determined that a sample size of 90 participants will have 80% power to detect an effect size of 0.30 (Cohen's D) using a paired t-test with a 0.05 two-sided significance level; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = .9789

3. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) - Rate at 2 Months Follow up
Description: Based on an interview with the participant, the clinician rates the total improvement on a 7 point scale as follows: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Time Frame: 2 months
Population: Nine participants did not participate in the clinicial interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 88
Participants
  CGI-I score of "1", "2" or "3" | 77
  CGI-I score of "4" or higher | 11

4. Secondary Outcome: Conners' Continuous Performance Test-3 (CPT-3) - Detectability (d') at Baseline and 2 Months Follow up
Description: Conners' Continuous Performance Test-3 (CPT-3) is an objective test of attention and impulsivity that has been validated in individuals aged 8 years and older.
  d-prime (d') is a measure of how well the respondent discriminates nontargets (i.e., the letter X) from targets (i.e., all other letters). This variable is also a signal detection statistic that measures the difference between the signal (targets) and noise (non-targets) distributions. In general, the greater the difference between the signal and noise distributions, the better the ability to distinguish non-targets and targets.
  CPT scores are age and gender standardized T-scores, in which the mean is equal to 50 and the standard deviation is equal to 10. d' is reverse-scored so that higher raw score and T-score values indicate worse performance (i.e., poorer discrimination). Atypical scores are higher than 60 indicating "elevated" to "very elevated" performance.
Time Frame: Baseline, 2 months
Population: Four participants did not complete the CPT.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Active
Number analyzed (Participants) | 93
T-score
  Baseline | 50.03 (0.90)
  End of Study | 47.95 (1.06)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.027, t-test, 2 sided; Mean Difference (Final Values) = 2.09

5. Secondary Outcome: Behavior Rating Inventory of Executive Function Adult Version (BRIEF-A) - Metacognitive Index - at Baseline and 2 Months Follow up
Description: The Behavior Rating Inventory of Executive Function Adult Version (BRIEF-A) is a standardized measure that captures views of adults' executive functions or self-regulation in their everyday environment. Items are rated on a 3-points Likert scale of 1 ('Never') to 3 ('Often').
  The Metacognition Index (MI) of the BRIEF-A reflects the individual's ability to initiate activity and generate problem-solving ideas, to sustain working memory, to plan and organize problem-solving approaches, to monitor success and failure in problem solving, and to organize one's materials and environment. The MI subscale includes 40-items with score ranges between 40 to 120. Higher values represent worse outcome and greater difficulties with executive functions.
Time Frame: Baseline, 2 months
Population: Four participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale (raw scores)
Arm/Group | Active
Number analyzed (Participants) | 93
score on a scale (raw scores)
  Baseline | 79.85 (1.75)
  End of Study | 77.76 (1.75)
Statistical Analysis 1: Comparison: Active; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.029, t-test, 2 sided; Mean Difference (Final Values) = 2.09

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the two-month intervention period.
Description: All side effects were transient, reported to be mild or moderate, and resolved after the removal of the glasses.
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 64/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=100)
Headache (General disorders) | 36
Eyestrain (General disorders) | 20
Dizziness (General disorders) | 18
Tiredness (General disorders) | 9
Discomfort (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT05777785/Prot_SAP_000.pdf